CLINICAL TRIAL: NCT05231538
Title: Effects of Neurodevelopment Therapy on Gross Motor Function and Postural Control in Children With Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Neurodevelopmental Therapy for Spastic Cerebral Palsy
Acronym: NDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Abdullah Khalid Khan, Principal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/882/2021
Record Dates: First submitted 2022-01-15; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Spastic; Diplegia, Spastic
Keywords: Neurodevelopmental therapy; NDT; Spastic cerebral palsy; Physical Therapy; Rehabilitation; Neurorehabilitation
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: Assessor was blind to treatment regimen administered to both groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental Therapy (Experimental): The treatment group received neurodevelopment treatment lasting for 3 months (3sessions per week). Additionally, for this study, the NDT programme included passive stretching of the lower limb muscles (e.g. hamstrings, gastrocsoleus), followed by techniques of reducing spasticity and facilitating more normal patterns of movement while working on motor functions. In each session, exercises included patients sustaining themselves on their forearms and hands, sitting, crawling, semi-kneeling, and in standing positions supported by the Physical therapist until tone reduction achieved. Balance and corrective reactions were developed by using a CP ball and tilt board.
  Interventions: Other: Neurodevelopmental therapy
- Routine Physical Therapy (Active Comparator): The control group underwent the exercises (stretching, passive range of motion, and active range of motion).
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Neurodevelopmental therapy — NDT is a hands-on, 'problem solving approach'. It is used in the management and treatment of children who have disorders of function, movement or postural control because of damage in their central nervous system.
  Arms: Neurodevelopmental Therapy
Other: Routine physical therapy — stretching, passive range of motion, and active range of motion).
  Arms: Routine Physical Therapy

SUMMARY:
This study was conducted to find out the Effects of Neurodevelopment therapy (a rehabilitative program designed by Bobath) on Gross Motor Function and Postural Control in Children with Spastic Cerebral Palsy. To investigate either there was a significant difference between the effects of neurodevelopment therapy and routine physical therapy on gross motor function and postural control in children with Spastic Cerebral Palsy.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted at Department of pediatric rehabilitation, Sher e Rabbani Hospital, Sheikhupura. Sample size was 66 and purposive sampling technique was adopted to collect data. Sample selection was completely based on inclusion and exclusion criteria. A diagnosed Spastic Cerebral Palsy patient aged 2-6 years with no other severe abnormalities such as seizure were recruited. While patients with mental retardation or undergone medical procedures likely to affect motor function such as botulinum toxin injections, orthopedic remedial surgery were excluded. Data was collected at baseline, 4th, 8th and 12th week of the treatment sessions. Gross motor function measure scale (GMFM-88) and posture and postural ability scale (PPAS) were used as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* • A diagnosed Spastic Cerebral Palsy (patient's diagnosis of CP confirmed by an expert pediatrician neurologist)

  * Spastic CP
  * No other severe abnormalities such as seizure
  * Aged 2-6 years
  * Both Genders

Exclusion Criteria:

* Medical procedures likely to affect motor function such as botulinum toxin injections
* Orthopedic remedial surgery
* Mental retardation, or a learning disability.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Scale (GMFS) | 12 weeks
  The Gross motor function scale (GMFS) is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring system of the GMFM is a four-point scale divided into five categories lying and rolling; sitting; crawling and kneeling; standing; walking, running
The Posture and Postural Ability Scale (PPAS) | 12 weeks
  The Posture and Postural Ability Scale (PPAS) is a 7-point ordinal scale for the assessment of postural ability in standing, sitting, supine and prone. There are six items for assessment of quality of posture in the frontal plane and another six items in the sagittal plane

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Khalid khan, MSNPT, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No